CLINICAL TRIAL: NCT03068988
Title: Mesenchymal Stem Cells in the Reconstruction Surgery of the Supraspinatus Muscle Lesions
Brief Title: Clinical Study on Mesenchymal Stem Cells Used in the Reconstruction Surgery of the Supraspinatus Muscle Lesions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Znojmo (Other)
Responsible Party: Principal Investigator, MUDr. Petr Šmíd, Prinicpal investigator, Doctor, Hospital Znojmo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016/05/25/09
Record Dates: First submitted 2017-02-20; First posted 2017-03-03 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Rotator Cuff Tear
Keywords: bone marrow stem cells; rotator cuff lesion
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mesenchymal stem cells (Experimental): mesenchymal stem cells concentrate into the supraspinatus footprint during the surgery
  Interventions: Biological: mesenchymal stem cells
- without mesenchymal stem cells (Placebo Comparator): rotator cuff surgery without mesenchymal stem cells
  Interventions: Procedure: without mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — mesenchymal stem cells concentrate into the supraspinatus footprint during the surgery
  Arms: mesenchymal stem cells
Procedure: without mesenchymal stem cells — rotator cuff surgery without mesenchymal stem cells
  Arms: without mesenchymal stem cells

SUMMARY:
The prospective randomized clinical study investigating the effect of mesenchymal stem cells on tendon healing. The objective of the study is to demonstrate the effect of concentrated bone marrow stem cells ( MSCs ) to the healing of sutured tendon of the supraspinatus muscle in comparison to the same procedure performed without MSCs. We have postulated the hypothesis that MSCs enhance the healing of the sutured supraspinatus tendon to its humeral footprint.

DETAILED DESCRIPTION:
The prospective randomized study is carried out at orthopaedic and traumatology, haematology and radiology departments. 50 patients were included in the study. Of the 25 patients in both groups, Group I (received the concentrate of marrow MSCs into the tendon- bone contact point at the site of the suture during surgery ) consisted of 7 women and 18 men ( mean age 51,2 years ), Group II ( without the use of MSCs ) consisted of 15 women and 10 men ( mean age 50,5 years ). Selection of patients into both groups was performed using permutation block randomization computer software Random Number Generator Software 7.0. All of radiographs/MRI/CT results were evaluated by an experienced radiologist specialized in musculoskeletal pathologies, that was blinded to the both groups of patients. Before entering the study, patients signed an informed consent created by the Ethical Committee of local hospital and were randomly assigned to one of the treatment possibilities with use of the Random Number Generator Software 7.0 by the method 1:1.

Before the surgical treatment, patients completed a questionnaire with VAS score, ASES score ( American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form ) and the Constant score. Further clinical control with completing these questionnaires is 6 months after surgery, 1 year after surgical treatment, 2, 5 and ten years postoperatively. Two years after the surgery MRI examination of the shoulder joint is performed. All of the outpatient clinical evaluations during the study were performed by the orthopaedic surgeon blinded to the both groups of patients.

The actual therapy was as follows: open surgery was preceded by a standard diagnostic arthroscopy, which was performed from the posterior portal for optics and anterior portal for arthroscopic instruments. The tendons of the rotator cuff were assessed from both sides - intraarticular and subacromial. To evaluate cuff tendon injury perioperatively and to measure the rupture width, a special arthroscopic hook calibrated in 1 mm was used. To evaluate the shape of the rupture, the classification of Ellman - Gartsman was used. Surgical treatment of injured tendons of the rotator cuff was performed in the beach chair position of the patient, by the deltoid muscle split approach. After evaluation of the extent and location of the cuff tendon lesion the aspiration of 10 ml of bone marrow blood was done ( from the humeral head through the same surgical approach ) into a 20 mL syringe prefilled with 0.5 ml of heparin with the Yamshidi needle. Aspiration of the bone marrow was performed by surgeon. From one bone puncture was aspirated maximally 3 ml of marrow blood. Centrifugation of the aspirate in 10 ml test-tube Monovette filled with citrate followed. Selected centrifugation regime consisted of gradient 15 minute centrifugation at 200 g RCF ( relative centrifugal force ). After such a centrifugation the tube contents is divided into three parts. The upper layer consists of the platelet-rich plasma (PRP), the middle layer of the buffy coat with the dominant proportion of leukocytes, and the lower layer is formed by sedimented erythrocytes. Using a sterile laboratory pipette, a collection of the buffy coat was performed. MSCs represented 0.01 to 0.02 % of all nuclear elements of the buffy coat, that is about 10 x 106 / l. The MSCs concentrate ( similar to synovial fluid in consistency and colour ) was impregnated into the collagen patch Hypro-Sorb F ( Otrokovice, Czech Republic ) of dimensions 1x2 cm. The collagen patch as a carrier of the MSCs concentrate was used to ensure its retention in desired place. This material was then inserted between the tendon and bone, into the place of re-fixing of the rotator cuff tendons ( footprint ) before tightening the threads of the anchors. Fixation of the tendon to the bone was made by a double row method with use of absorbable fixation anchors BioComposite Corkscrew ( Arthrex, Munich, Germany ). In all such treated cases the tendon was fixed in place of original attachment without any stress and without the need of abduction of the arm above 60 degrees. All patients underwent Neer acromioplasty for an increase of the subacromial space. This procedure was followed by the standard surgical wound closure in all anatomical layers, sterile dressing of the wound and by applying of the abduction orthosis. All patients were operated by the same orthopaedic surgeon with the same surgical technique. Open surgery instead of arthroscopy was chosen because of the safer fixation of the MSCs carrier under the re-inserted tendon and to reduce the risk of washout of the MSCs concentrate from the carrier during the arthroscopy.

Surgical treatment of patients in Group II was identical as in Group I, except the aspiration of bone marrow from the humeral head and subsequent application of the scaffold saturated with MSCs into the tendon / bone interface.

Abduction fixation lasted for 4 weeks. Passive motion over the horizontal line under the guidance of a physiotherapeutist was initiated the first postoperative day. After removing the fixation, an active rehabilitation began, that is a full range of motion exercises done actively 6 weeks after surgery. Full load was allowed 12 weeks after the surgery.

Outpatient follow-up took place according to the schedule mentioned above. To check the integrity of the tendon at the point of insertion into the greater tuberosity of the humerus, MRI of the shoulder joint was performed 2 years postoperatively. Both, preoperative and postoperative MRI examinations were performed with a 1.5T high-field scanner, in sagittal, coronal, and axial planes, in T1- and T2-weighted fat-saturated sequences ( MRI arthrography using gadollinium as a contrast medium ). All of MRI results were evaluated by an experienced radiologist specialized in musculoskeletal pathologies. He evaluated tendon integrity, presence and localisation of complete retear, tendon and muscle borders, and presence of abnormal artifacts.

The primary hypothesis of this study is that the use of mesenchymal stem cells in the supraspinatus tendon reconstruction surgery will have a positive effect in the assessment of both subjective and objective scoring systems, and also in terms of reducing the number of tendon reruptures compared to the patients population in which mesenchymal stem cells were not used. All data were statistically analyzed with STATISTICA 9.0 programme. To compare the results of the of the VAS score, the Constant score, and the ASES score preoperatively and one year after the surgery Student´s t- test was used, to compare the incidence of reruptures between both groups of patients 2 years postoperatively Chi-square test was used. The significance level was determined at p <0.05. Patients were randomly assigned to one of the treatment possibilities with use of the Random Number Generator Software 7.0 by the method 1:1

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18-60 years
* chronic supraspinatus tendon tear greater than 50% of its width
* no history of trauma to the examined shoulder girdle
* confirmation by the clinical examination and preoperative imaging examination ( MRI arthrography )
* signed informed consent
* minimum preoperative haemoglobin concentration in men 13.8 g / dl, in women 12.1 g / dl

Exclusion Criteria:

* previous surgical treatment of the rotator cuff
* cuff tear arthropathy grade 3-5 according to Hamada
* fatty degeneration of the cuff muscle ( Goutallier 3 and 4 )
* atrophy of the supraspinatus muscle according to the Thomazeau classification grade II and III
* retraction of the supraspinatus muscle tendon Patte III
* pregnancy
* active infection at the surgical site or elsewhere in the body
* osteomyelitis
* sepsis
* history of diabetes
* steroids use
* chemotherapy
* use of NSAIDs
* radiation
* hepatitis
* HIV
* hemato / oncological diseases
* alcohol abuse
* drug abuse
* cigarettes
* medical condition that affects the growth of bone or connective tissue (osteomalacia or other metabolic bone disease)
* vascular insufficiency
* operated extremity muscle atrophy
* neuromuscular disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The supraspinatus tendon re-rupture rate | 2 years postoperatively
  presence of the supraspinatus tendon rupture on magnetic resonance imaging evaluated 2 years after the surgery, incidence of rerupture compared between group I- with the use of mesenchymal stem cells and group II- without the use of mesenchymal stem cells

SECONDARY OUTCOMES:
visual analogue scale | 1 day before the surgery, 6 months postoperatively, 1 year postoperatively, 2 years postoperatively, 5 years postoperatively, 10 years postoperatively
  patients subjectively rate the pain level at 6 grade scale from 0-5 where 0 represents no pain and 5 excruciating pain
ASES score- American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form | 1 day before the surgery, 6 months postoperatively, 1 year postoperatively, 2 years postoperatively, 5 years postoperatively, 10 years postoperatively
  Consists of two parts. The first part features a questionnaire filled in by the patients themselves, and included a visual analogue scale for pain and instability and assessment of ability to perform activities of daily living ( ADL ). The second part, which is completed by a doctor, represents an objective assessment of the conditions, and includes the evaluation of range of motion, specific physical characteristics, strength and stability. Score for the arm was then derived from the visual analogue scale for pain (50%) and the general score for ADL (50%).
Constant score | 1 day before the surgery, 6 months postoperatively, 1 year postoperatively, 2 years postoperatively, 5 years postoperatively, 10 years postoperatively
  Two parts: first- subjective evaluation of ADL ( activities of daily living ) from the patient's perspective, the second part is an objective assessment of range of motion and muscle strength performed by the physician

CONTACTS AND LOCATIONS:
Overall Officials: Petr Šmíd, Dr., Principal Investigator — General Hospital Znojmo, Czech Republic
Locations (1):
- Petr Šmíd, Znojmo, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goutallier D, Postel JM, Bernageau J, Lavau L, Voisin MC. Fatty muscle degeneration in cuff ruptures. Pre- and postoperative evaluation by CT scan. Clin Orthop Relat Res. 1994 Jul;(304):78-83. PMID 8020238
- [Result] Thomazeau H, Boukobza E, Morcet N, Chaperon J, Langlais F. Prediction of rotator cuff repair results by magnetic resonance imaging. Clin Orthop Relat Res. 1997 Nov;(344):275-83. PMID 9372778
- [Result] Patte D. Classification of rotator cuff lesions. Clin Orthop Relat Res. 1990 May;(254):81-6. PMID 2323151
- [Result] Richards RR, An KN, Bigliani LU, Friedman RJ, Gartsman GM, Gristina AG, Iannotti JP, Mow VC, Sidles JA, Zuckerman JD. A standardized method for the assessment of shoulder function. J Shoulder Elbow Surg. 1994 Nov;3(6):347-52. doi: 10.1016/S1058-2746(09)80019-0. Epub 2009 Feb 13. PMID 22958838
- [Result] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738